CLINICAL TRIAL: NCT00730171
Title: An Open-label, Long-term Safety Study of Oral Linaclotide Administered to Patients With Chronic Constipation or Irritable Bowel Syndrome With Constipation
Brief Title: An Open-label, Long-term Safety Study of Linaclotide in Patients With Chronic Constipation or Irritable Bowel Syndrome With Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ironwood Pharmaceuticals, Inc. (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCP-103-305
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-01

CONDITIONS: Irritable Bowel Syndrome With Constipation; Chronic Constipation
MeSH Terms: interventions — linaclotide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

ARMS (1):
- Linaclotide (Experimental): Linaclotide 290 μg/day capsules, administered orally once daily for up to 78 weeks. Dose reduction to 145 μg/day was permitted at the discretion of the Investigator.
  Interventions: Drug: Linaclotide

INTERVENTIONS:
Drug: Linaclotide — Linaclotide capsules, oral, once daily each morning at least 30 minutes before breakfast for the duration of the study.
  Other Names: Linzess

SUMMARY:
The objective of this study is to assess the long-term safety of linaclotide administered to patients with chronic constipation (CC) or irritable bowel syndrome with constipation (IBS-C).

DETAILED DESCRIPTION:
Participants include randomization-ineligible (RI) patients from the lead-in double-blind trials MCP-103-302 (NCT00938717) or MCP-103-303 (NCT00730015), or rollover (RO) patients from the lead-in double-blind trials MCP-103-302 (NCT00938717), MCP-103-303 (NCT00730015), and from the Phase 2 double-blind studies MCP-103-004 (NCT00306748), MCP-103-005 (NCT00258193), and MCP-103-201 (NCT00402337), or MCP-103-202 (NCT00460811).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have

  * entered study MCP-103-303 or MCP-103-302 and at minimum completed the pre-treatment period or
  * completed one of the following studies: MCP-103-004, MCP-103-005, MCP-103-201, MCP-103-202
* Sexually active patients of childbearing potential agree to use birth control
* Females of childbearing potential must have a negative urine pregnancy test prior to dosing
* Lactating females must agree not to breastfeed
* Patient must meet protocol criteria for CC or IBS-C

Exclusion Criteria:

* Patient must not use protocol-defined prohibited medicine
* Patient is planning to receive an investigational drug at any time during the study
* Patient has an unresolved adverse events or a clinically significant finding on a physical examination, 12-lead electrocardiogram, or clinical laboratory test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1743 (Actual)
Dates: Start 2008-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M. Johnston, MD, FACP, Study Chair — Ironwood Pharmaceuticals, Inc.
Locations (109):
- United States (109):
  - Ironwood Investigational Site, Birmingham, Alabama
  - Ironwood Investigational Site, Huntsville, Alabama
  - Ironwood Investigational Site, Chandler, Arizona
  - Ironwood Investigational Site, Phoenix, Arizona
  - Ironwood Investigational Site, Tucson, Arizona
  - Ironwood Investigational Site, Sherwood, Arkansas
  - Ironwood Investigational Site, Anaheim, California
  - Ironwood Investigational Site, Chula Vista, California
  - Ironwood Investigational Site, Encinitas, California
  - Ironwood Investigational Site, Garden Grove, California
  - Ironwood Investigational Site, Laguna Hills, California
  - Ironwood Investigational Site, Los Angeles, California
  - Ironwood Investigational Site, Orange, California
  - Ironwood Investigational Site, Sacramento, California
  - Ironwood Investigational Site, San Carlos, California
  - Ironwood Investigational Site, San Diego, California
  - Ironwood Investigational Site, Colorado Springs, Colorado
  - Ironwood Investigational Site, Bristol, Connecticut
  - Ironwood Investigational Site, Boynton Beach, Florida
  - Ironwood Investigational Site, Hollywood, Florida
  - Ironwood Investigational Site, Inverness, Florida
  - Ironwood Investigational Site, Jacksonville, Florida
  - Ironwood Investigational Site, Lauderdale Lakes, Florida
  - Ironwood Investigational Site, Miami, Florida
  - Ironwood Investigational Site, Pinellas Park, Florida
  - Ironwood Investigational Site, Port Orange, Florida
  - Ironwood Investigational Site, Tampa, Florida
  - Ironwood Investigational Site, Newnan, Georgia
  - Ironwood Investigational Site, Peoria, Illinois
  - Ironwood Investigational Site, Anderson, Indiana
  - Ironwood Investigational Site, Clive, Iowa
  - Ironwood Investigational Site, Davenport, Iowa
  - Ironwood Investigational Site, Mission, Kansas
  - Ironwood Investigational Site, Overland Park, Kansas
  - Ironwood Investigational Site, Topeka, Kansas
  - Ironwood Investigational Site, Baton Rouge, Louisiana
  - Ironwood Investigational Site, Metairie, Louisiana
  - Ironwood Investigational Site, Monroe, Louisiana
  - Ironwood Investigational Site, Shreveport, Louisiana
  - Ironwood Investigational Site, Annapolis, Maryland
  - Ironwood Investigational Site, Baltimore, Maryland
  - Ironwood Investigational Site, Hollywood, Maryland
  - Ironwood Investigational Site, Laurel, Maryland
  - Ironwood Investigational Site, Chesterfield, Michigan
  - Ironwood Investigational Site, Traverse City, Michigan
  - Ironwood Investigational Site, Troy, Michigan
  - Ironwood Investigational Site, Plymouth, Minnesota
  - Ironwood Investigational Site, Jackson, Mississippi
  - Ironwood Investigational Site, Tupelo, Mississippi
  - Ironwood Investigational Site, Jefferson City, Missouri
  - Ironwood Investigational Site, Henderson, Nevada
  - Ironwood Investigational Site, Las Vegas, Nevada
  - Ironwood Investigational Site, Cedar Knolls, New Jersey
  - Ironwood Investigational Site, Marlton, New Jersey
  - Ironwood Investigational Site, Ocean City, New Jersey
  - Ironwood Investigational Site, Albuquerque, New Mexico
  - Ironwood Investigational Site, Mineola, New York
  - Ironwood Investigational Site, Pittsford, New York
  - Ironwood Investigational Site, Asheboro, North Carolina
  - Ironwood Investigational Site, Asheville, North Carolina
  - Ironwood Investigational Site, Chapel Hill, North Carolina
  - Ironwood Investigational Site, Charlotte, North Carolina
  - Ironwood Investigational Site, Greensboro, North Carolina
  - Ironwood Investigational Site, Harrisburg, North Carolina
  - Ironwood Investigational Site, Hickory, North Carolina
  - Ironwood Investigational Site, Huntersville, North Carolina
  - Ironwood Investigational Site, Jacksonville, North Carolina
  - Ironwood Investigational Site, New Bern, North Carolina
  - Ironwood Investigational Site, Statesville, North Carolina
  - Ironwood Investigational Site, Summerville, North Carolina
  - Ironwood Investigational Site, Wilmington, North Carolina
  - Ironwood Investigational Site, Winston-Salem, North Carolina
  - Ironwood Investigational Site, Beachwood, Ohio
  - Ironwood Investigational Site, Cincinnati, Ohio
  - Ironwood Investigational Site, Dayton, Ohio
  - Ironwood Investigational Site, Mentor, Ohio
  - Ironwood Investigational Site, Sylvania, Ohio
  - Ironwood Investigational Site, Wadsworth, Ohio
  - Ironwood Investigational Site, Zanesville, Ohio
  - Ironwood Investigational Site, Oklahoma City, Oklahoma
  - Ironwood Investigational Site, Yukon, Oklahoma
  - Ironwood Investigational Site, Lancaster, Pennsylvania
  - Ironwood Investigational Site, Levittown, Pennsylvania
  - Ironwood Investigational Site, Pittsburgh, Pennsylvania
  - Ironwood Investigational Site, Sellersville, Pennsylvania
  - Ironwood Investigational Site, Anderson, South Carolina
  - Ironwood Investigational Site, Charleston, South Carolina
  - Ironwood Investigational Site, Simpsonville, South Carolina
  - Ironwood Investigational Site, Bristol, Tennessee
  - Ironwood Investigational Site, Chattanooga, Tennessee
  - Ironwood Investigational Site, Germantown, Tennessee
  - Ironwood Investigational Site, Kingsport, Tennessee
  - Ironwood Investigational Site, Nashville, Tennessee
  - Ironwood Investigational Site, Beaumont, Texas
  - Ironwood Investigational Site, El Paso, Texas
  - Ironwood Investigational Site, Fort Worth, Texas
  - Ironwood Investigational Site, Houston, Texas
  - Ironwood Investigational Site, Irving, Texas
  - Ironwood Investigational Site, Longview, Texas
  - Ironwood Investigational Site, San Antonio, Texas
  - Ironwood Investigational Site, Sugar Land, Texas
  - Ironwood Investigational Site, Ogden, Utah
  - Ironwood Investigational Site, Salt Lake City, Utah
  - Ironwood Investigational Site, Chesapeake, Virginia
  - Ironwood Investigational Site, Lynchburg, Virginia
  - Ironwood Investigational Site, Spokane, Washington
  - Ironwood Investigational Site, Vancouver, Washington
  - Ironwood Investigational Site, La Crosse, Wisconsin
  - Ironwood Investigational Site, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were categorized as either randomization-ineligible (RI) from the lead-in double-blind trials MCP-103-302 or MCP-103-303, or rollover (RO) from lead-in double-blind trials MCP-103-302, MCP-103-303, and from Phase 2 double-blind studies MCP-103-004, MCP-103-005, and MCP-103-201, or MCP-103-202 (See Detailed Description for NCT numbers).
Pre-assignment Details: A total of 1743 participants were enrolled in the study; 1725 received ≥1 dose of open-label linaclotide (included in the Overall Safety Population). One participant enrolled twice in the study under 2 ID numbers and is included as an RI participant in the CC Safety Population, and as an RO participant in the IBS-C and Overall Safety Populations.
Groups:
- Overal Safey Population: Total: All RI and RO participants who received linaclotide 290 μg/day capsules, administered orally once daily for up to 78 weeks. Dose reduction to 145 μg/day was permitted at the discretion of the Investigator if a participant experienced AEs intolerable enough to prompt consideration of study withdrawal. After a temporary suspension of dosing, participants may have received either 145 μg/day or 290 μg/day of linaclotide, at the discretion of the Investigator. Subsequent dose adjustments (increases or decreases between 290 μg/day and 145 μg/day) were permitted also at the Investigator's discretion.
Period: Overall Study
Arm/Group | Overal Safey Population: Total
Started | 1725
CC Safety Population (met the modified Rome II criteria for chronic constipation (CC)) | 607
IBS-C Safety Population (met the modified Rome II criteria for irritable bowel syndrome with constipation (IBS-C)) | 1119
Completed | 954
Not Completed | 771
Not completed — Didn't Meet Inclusion/Exclusion Criteria | 5
Not completed — Adverse Event | 193
Not completed — Protocol Violation | 48
Not completed — Withdrawal by Subject | 202
Not completed — Lost to Follow-up | 121
Not completed — Insufficient Therapeutic Response | 141
Not completed — Other | 61

BASELINE CHARACTERISTICS:
Population: Overall Safety Population: enrolled participants who received at least 1 dose of open-label study drug.
Groups:
- Overall Safety Population: All RI and RO participants who received linaclotide 290 μg/day capsules, administered orally once daily for up to 78 weeks. Dose reduction to 145 μg/day was permitted at the discretion of the Investigator if a participant experienced AEs intolerable enough to prompt consideration of study withdrawal. After a temporary suspension of dosing, participants may have received either 145 μg/day or 290 μg/day of linaclotide, at the discretion of the Investigator. Subsequent dose adjustments (increases or decreases between 290 μg/day and 145 μg/day) were permitted also at the Investigator's discretion.
Arm/Group | Overall Safety Population
Number analyzed (Participants) | 1725
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1532
  Male | 193

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Treatment-Emergent Adverse Event (TEAE)
Description: For RI and Phase 2 RO participants, an AE that occurred during the study was considered a TEAE if it was not present before the day of the first dose of open-label study drug, or was present before the day of the first dose of open-label study drug but increased in severity on or after that day. For Phase 3 RO participants, an AE that occurred during the study was considered a TEAE if it was not present before the day of the first dose of double-blind study drug in trial MCP-103-302 or MCP-103-303, or was present before the day of the first dose of double-blind study drug in those trials but increased in severity on or after that day. Deaths and serious AEs (SAEs) are those that occurred on or after the date of the first dose of open-label study drug, and within 30 days of the date of last dose of open-label study drug.
Time Frame: From first dose of open-label study drug up to 78 weeks
Population: Enrolled participants who received at least 1 dose of open-label study drug. It was identified that 1 participant enrolled twice in the study under 2 ID numbers; this participant is included as an RI participant in the CC Safety Population, and as an RO participant in both the IBS-C and Overall Safety Populations.
Measure: Count of Participants; unit: Participants
Groups:
- CC Safety Population: Total: RI and RO participants who met the Rome II criteria for CC and who received linaclotide 290 μg/day capsules, administered orally once daily for up to 78 weeks. Dose reduction to 145 μg/day was permitted at the discretion of the Investigator.
- IBS-C Safety Population: Total: RI and RO participants who met the Rome II criteria for IBS-C and who received linaclotide 290 μg/day capsules, administered orally once daily for up to 78 weeks. Dose reduction to 145 μg/day was permitted at the discretion of the Investigator.
- Overall Safety Population: Total: All RI and RO participants who received linaclotide 290 μg/day capsules, administered orally once daily for up to 78 weeks. Dose reduction to 145 μg/day was permitted at the discretion of the Investigator.
Arm/Group | CC Safety Population: Total | IBS-C Safety Population: Total | Overall Safety Population: Total
Number analyzed (Participants) | 607 | 1119 | 1725
Participants | 65 | 389 | 454

ADVERSE EVENTS:
Time Frame: From first dose of open-label study drug up to 78 weeks for adverse events (AEs) and within 30 days of last dose of study drug (up to 82 weeks) for serious AEs.
Description: It was identified that 1 participant enrolled twice in the study under 2 ID numbers; this participant is included as an RI participant in the CC Safety Population, and as an RO participant in both the IBS-C and Overall Safety Populations.
Groups:
- CC Safety Population: Total: RI and RO participants who met the modified Rome II criteria for CC and who received linaclotide 290 μg/day capsules, administered orally once daily for up to 78 weeks. Dose reduction to 145 μg/day was permitted at the discretion of the Investigator.
- IBS-C Safety Population: Total: RI and RO participants who met the modified Rome II criteria for IBS-C and who received linaclotide 290 μg/day capsules, administered orally once daily for up to 78 weeks. Dose reduction to 145 μg/day was permitted at the discretion of the Investigator.
Arm/Group | CC Safety Population: Total | IBS-C Safety Population: Total | Overall Safety Population: Total
All-Cause Mortality (participants affected / at risk) | 2/607 | 2/1119 | 4/1725
Serious Adverse Events (participants affected / at risk) | 41/607 | 56/1119 | 97/1725
Other Adverse Events (participants affected / at risk) | 283/607 | 572/1119 | 855/1725
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CC Safety Population: Total (N=607) | IBS-C Safety Population: Total (N=1119) | Overall Safety Population: Total (N=1725)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 3 | 6
Acute myocardial infarction (Cardiac disorders) | 2 | 1 | 3
Bradycardia (Cardiac disorders) | 2 | 0 | 2
Cystocele (Reproductive system and breast disorders) | 2 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 2
Diverticular perforation (Gastrointestinal disorders) | 2 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 2
Adenomyosis (Reproductive system and breast disorders) | 1 | 0 | 1
Aplastic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Bipolar I disorder (Psychiatric disorders) | 1 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 4
Chest pain (General disorders) | 1 | 1 | 2
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 1 | 2
Convulsion (Nervous system disorders) | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 2 | 3
Depression (Psychiatric disorders) | 1 | 2 | 3
Diverticulitis (Gastrointestinal disorders) | 1 | 1 | 2
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 1 | 2
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 1
Endometrial hypertrophy (Reproductive system and breast disorders) | 1 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 3
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Malocclusion (Gastrointestinal disorders) | 1 | 0 | 1
Micrognathia (Congenital, familial and genetic disorders) | 1 | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 1
Oesophageal squamous cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Peritonitis (Gastrointestinal disorders) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2 | 3
Pneumothorax traumatic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Prognathism (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Rectocele (Reproductive system and breast disorders) | 1 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 1
Thyrotoxic crisis (Endocrine disorders) | 1 | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 1 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 3 | 3
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 2 | 2
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 2 | 2
Bronchitis (Infections and infestations) | 0 | 2 | 2
Gastroenteritis (Infections and infestations) | 0 | 2 | 2
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 1
Anorexia nervosa (Psychiatric disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 1
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 1
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 1
Clostridial infection (Infections and infestations) | 0 | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 1 | 1
Gastroenteritis salmonella (Infections and infestations) | 0 | 1 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypothermia (General disorders) | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 1
Intertrigo candida (Infections and infestations) | 0 | 1 | 1
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 1 | 1
Meningitis viral (Infections and infestations) | 0 | 1 | 1
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 1
Oedema peripheral (General disorders) | 0 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CC Safety Population: Total (N=607) | IBS-C Safety Population: Total (N=1119) | Overall Safety Population: Total (N=1725)
Diarrhoea (Gastrointestinal disorders) | 179 | 358 | 537
Abdominal pain (Gastrointestinal disorders) | 23 | 74 | 97
Nausea (Gastrointestinal disorders) | 36 | 59 | 95
Constipation (Gastrointestinal disorders) | 16 | 65 | 81
Flatulence (Gastrointestinal disorders) | 34 | 36 | 70
Urinary tract infection (Infections and infestations) | 44 | 85 | 129
Sinusitis (Infections and infestations) | 40 | 83 | 123
Upper respiratory tract infection (Infections and infestations) | 27 | 61 | 88

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may publish or disclose the results of the study 24 months after final data lock provided that sponsor can review the publication prior to public release, sponsor can request removal of confidential information of sponsor (not including results of trial), and sponsor can request a publication delay in order to protect potentially patentable information. Furthermore, if a publication committee is developing an initial publication, PI is to delay disclosure until that publication is published